CLINICAL TRIAL: NCT03495609
Title: The Use of Recombinant hCG to Prevent Breast Cancer in BRCA1 and BRCA2 Carriers
Brief Title: Use of Recombinant hCG to Prevent Breast Cancer in BRCA1 and BRCA2 Carriers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Fox Chase Cancer Center (Other); Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-001720-36
Record Dates: First submitted 2018-01-23; First posted 2018-04-12 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: hCG; BRCA1 Mutation; BRCA2 Mutation
MeSH Terms: interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovitrelle (Experimental)
  Interventions: Drug: Ovitrelle

INTERVENTIONS:
Drug: Ovitrelle — Ovitrelle will be injected in 35 asymptomatic women with BRCA1 or BRCA2 mutation during 90 days (an extra 4 weeks in a subgroup). The gene expression of the breast epithelial cells will be characterized and compared to the gene expression of the breast epithelial cells before ovitrelle injection.

SUMMARY:
Specific aim: To establish the proof of principle that treatment of "high breast cancer risk" women with recombinant human chorionic gonadotropin (r-hCG) will change their breast epithelium's high risk genomic profile to one similar to that identified in women with a history of early full first term pregnancy.

DETAILED DESCRIPTION:
This study is based on the investigators preclinical data that have demonstrated that r-hCG exerts a mammary cancer preventive effect that is mediated by the induction of gland differentiation, which results in permanent changes in the genomic signature of this organ. This exploratory study will evaluate the genomic profile of breast epithelial cells obtained from random periareolar fine needle aspiration (RPFNA) specimens performed in high risk women treated for 90 days (an extra 4 weeks in a subgroup) with r-hCG. This knowledge will serve as the basis for establishing a novel genomic biomarker that will serve as a surrogate endpoint in future preventive clinical trials.

The objective of the proposed study is to characterize the genomic profile of breast epithelial cells obtained from 35 asymptomatic high breast cancer risk nulliparous premenopausal women carriers of BRCA1 and BRCA2 deleterious mutations. Gene expression measurements and benign breast tissue specimens will be obtained at baseline (time 0), after treatment with r-hCG at 90 days (time 1), at 270 days from baseline (time 2) and (in a subgroup) at 60 weeks (+/- 4 weeks).

The primary objective of the study is to compare the gene expression profiles of these women across the three (or four) time points and identify differentially expressed genes. The investigator is interested in comparing the expression profiles between all pairs of time points as well as across time. The comparison of profiles before and after treatment with r-hCG, both at 90 and 270 days are of particular interest. The women will receive 3x/week injections of 250 microgram r-hCG for a total of 12 weeks (an extra 4 weeks in a subgroup). Core Needle Biopsies specimens will be primarily utilized for analysis of genomic expression by cDNA microarray. In addition, a series of surrogate intermediate markers such as cytomorphologic evaluation and cell proliferation index will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal women
* BRCA1 carrier

Exclusion Criteria:

* History of allergic reaction to compounds of similar chemical or biologic composition to hCG
* receiving medication that could interfere with the study protocol objectives (hormonal contraceptives, androgens, prednisone, thyroid hormones, insulin)
* previous treatment with follicle stimulating hormone for assisted reproduction
* uncontrolled intercurrent illness
* Heart disease
* Severe cognitive decline
* Psychiatric desease
* HIV positive
* Hepatitis B or C infection

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only females who are BRCA1 or BRCA2 carriers and who are premenopausal will be included
Enrollment: 33 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Does Ovitrelle result in early prevention of breast cancer in BRCA1 and BRCA2 carriers? | 48 weeks
  The investigators are expecting that r-hCG is inducing genomic signature of protection in the breast. Participants will receive a subcutaneous injection of recombinant hCG three times a week for 12 (or 16) weeks. Normal breast tissue specimens will be collected by Spirotome at the beginning of treatment (day 0), at the end of treatment (week 13) and at 36 weeks. The specimens will be primarily utilized for analysis of genomic expression by cDNA microarray, RNA sequencing and epigenomic studies. In addition, a series of surrogate intermediate markers such as cytomorphologic evaluation and cell proliferation index will be analyzed. The primary objective is to compare the gene expression, and epigenomic profiles of sampled breast epithelial cells across the three time points and identify differentially expressed or silenced genes.

SECONDARY OUTCOMES:
Does Ovitrelle result in early prevention of breast cancer in BRCA1 and BRCA2 carriers? | 60 weeks
  The investigators are expecting that r-hCG is inducing genomic signature of protection in the breast. Participants will receive a subcutaneous injection of recombinant hCG three times a week for 12 (or 16) weeks. Normal breast tissue specimens will be collected by Spirotome at the beginning of treatment (day 0), at the end of treatment (week 13) and at 36 weeks. The specimens will be primarily utilized for analysis of genomic expression by cDNA microarray, RNA sequencing and epigenomic studies. In addition, a series of surrogate intermediate markers such as cytomorphologic evaluation and cell proliferation index will be analyzed. The primary objective is to compare the gene expression, and epigenomic profiles of sampled breast epithelial cells across the three time points and identify differentially expressed or silenced genes.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Russo, Prof., Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Ghent University Hospital, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No